CLINICAL TRIAL: NCT00116844
Title: Valacyclovir for the Suppression of HSV-2 Viral Shedding in HSV-2 Seropositive Individuals With No History of Symptomatic GH
Brief Title: VALTREX Once Daily For Viral Shedding In Herpes Simplex Virus 2 (HSV-2) Seropositive Subjects. VALTREX® Tablet is a Trademark of GlaxoSmithKline Group of Companies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VLX103596; NCT00268190 (obsolete NCT alias)
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-08

CONDITIONS: Infections, Herpesviridae
Keywords: viral shedding; Recurrent; herpes; genital herpes
MeSH Terms: conditions — Herpesviridae Infections; Recurrence; Herpes Simplex; Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: VALTREX 1 g once daily, Placebo (Experimental): VALTREX 1 g once daily, Placebo
  Interventions: Drug: Valaciclovir; Drug: Placebo
- Sequence 2: Placebo, VALTREX 1 g once daily (Experimental): Placebo, VALTREX 1 g once daily
  Interventions: Drug: Valaciclovir; Drug: Placebo

INTERVENTIONS:
Drug: Valaciclovir — Valtrex 1g once daily
Drug: Placebo — placebo

SUMMARY:
Eligible subjects will be randomized to receive VALTREX® tablet 1g or placebo once daily for 60 days in a two-way crossover study with a washout period of 7 days between treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* In overall general good health.
* HSV-2 (Herpes Simplex Virus-2) seropositive at screening.

Exclusion criteria:

* have active lesions consistent with genital herpes.
* previous history of symptomatic genital herpes.
* history of recurrent, undiagnosed symptoms consistent with genital herpes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-03-29 (Actual); Primary Completion 2006-01-10 (Actual); Study Completion 2006-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Davis, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: VLX103596 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March-2005 to January-2006, 73 participants from 13 centers in the United States were randomized into the study (36 in VALTREX™-Placebo, and 37 in Placebo-VALTEX treatment sequence). One participant in each treatment sequence did not receive study medication and intent-to-treat exposed (ITTE) population was comprised of 71 participants.
Pre-assignment Details: Eligible male or female immunocompetent participants in general good health were enrolled. Additionally, participants must be Herpes Simplex Virus Type 2 (HSV-2) seropositive at screening. VALTREX (valacyclovir hydrochloride) is registered trademark of GlaxoSmithKline.
Groups:
- Sequence 1: VALTREX 1 g Once Daily, Placebo: Participants randomized to this sequence received VALTREX 1 gram (g) once daily for 60 days, to be taken as two 500 milligram (mg) caplets in Period 1 followed by matching placebo for 60 days in Period 2 with 7 days of washout period between 2 periods. Participants were instructed to take caplets at approximately the same time of day each day, without regard to meals. If a dose was missed, the participants take the dose later that day provided they take it at least 2 hours before their next scheduled dose; otherwise the dose was omitted.
- Sequence 2: Placebo, VALTREX 1 g Once Daily: Participants randomized to this sequence received matching placebo for 60 days, to be taken as two 500 mg caplets in Period 1 followed by VALTREX 1 g once daily for 60 days in Period 2 with 7 days of washout period between 2 periods. Participants were instructed to take caplets at approximately the same time of day each day, without regard to meals. If a dose was missed, the participants take the dose later that day provided they take it at least 2 hours before their next scheduled dose; otherwise the dose was omitted.
Period: Period 1: Treatment Period 1 (60 Days)
Arm/Group | Sequence 1: VALTREX 1 g Once Daily, Placebo | Sequence 2: Placebo, VALTREX 1 g Once Daily
Started | 35 | 36
Completed | 28 | 33
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Other | 1 | 1
Period: Period 2: Washout Period (7 Days)
Arm/Group | Sequence 1: VALTREX 1 g Once Daily, Placebo | Sequence 2: Placebo, VALTREX 1 g Once Daily
Started | 28 | 33
Completed | 28 | 33
Not Completed | 0 | 0
Period: Period 1: Treatment Period 2 (60 Days)
Arm/Group | Sequence 1: VALTREX 1 g Once Daily, Placebo | Sequence 2: Placebo, VALTREX 1 g Once Daily
Started | 28 | 33
Completed | 24 | 28
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The ITTE population was defined as consisting of all participants who received at least one dose of investigational product and at least one safety and/or efficacy evaluation.
Groups:
- Sequence 1: VALTREX 1 g Once Daily, Placebo: Participants randomized to this sequence received VALTREX 1 g once daily for 60 days, to be taken as two 500 mg caplets in Period 1 followed by matching placebo for 60 days in Period 2 with 7 days of washout period between 2 periods. Participants were instructed to take caplets at approximately the same time of day each day, without regard to meals. If a dose was missed, the participants take the dose later that day provided they take it at least 2 hours before their next scheduled dose; otherwise the dose was omitted.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: VALTREX 1 g Once Daily, Placebo | Sequence 2: Placebo, VALTREX 1 g Once Daily | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (12.96) | 35.8 (11.69) | 37.4 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 14 | 19
  White | 28 | 19 | 47
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Days of Subclinical Shedding as Determined by Type-specific Polymerase Chain Reaction (PCR) Assay for HSV-2
Description: Percent of subclinical days with HSV-2 shedding was defined for each participant as the percent of subclinical days with PCR data for which HSV-2 shedding was detected by a positive PCR result, that is, the number of subclinical days with HSV-2 PCR shedding divided by total number of subclinical days with PCR data, multiplied by 100. For each participant, each study day was classified by PCR as 'shedding' or 'no shedding'; additionally each day was classified as 'clinical' (presence of genital lesions) or subclinical (no genital lesions). Genital/anal-rectal swabs was collected daily during each entire 60-day treatment period of each period and the washout period.
Time Frame: Up to Day 60 of each treatment period (up to 160 days)
Population: The intent-to-treat crossover (ITTC) population was defined as consisting of all participants who received at least one dose of investigational product and had at least one PCR swabbing result in each treatment period. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Groups:
- VALTREX 1 g Once Daily: Participants randomized to this arm received VALTREX 1g once daily for 60 days, to be taken as two 500 mg caplets in a two-way crossover design. Participants were instructed to take caplets at approximately the same time of day each day, without regard to meals. If a dose was missed, the participants take the dose later that day provided they take it at least 2 hours before their next scheduled dose; otherwise the dose was omitted. There was a washout period of seven days between treatment periods.
- Placebo: Participants randomized to this arm received matching placebo once daily for 60 days, to be taken as two caplets in a two-way crossover design. Participants were instructed to take caplets at approximately the same time of day each day, without regard to meals. If a dose was missed, the participants take the dose later that day provided they take it at least 2 hours before their next scheduled dose; otherwise the dose was omitted. There was a washout period of seven days between treatment periods.
Arm/Group | VALTREX 1 g Once Daily | Placebo
Number analyzed (Participants) | 56 | 56
Percentage of days | 1.5 (5.3) | 5.1 (9)
Statistical Analysis 1: Comparison: VALTREX 1 g Once Daily vs Placebo; Test type: Superiority or Other; p < 0.001, Nonparametric tests-Wilcoxon Rank Sum

2. Secondary Outcome: Mean Percent Days of Total HSV-2 Shedding
Description: The percent of days with total (clinical and subclinical) HSV-2 shedding was defined as the percent of all days with PCR data for which HSV-2 shedding was detected. Mean percent of days with total HSV-2 shedding was the statistic used to summarize this endpoint for each treatment group. For each participant, each study day was classified by PCR as 'shedding' or 'no shedding'; additionally each day was classified as 'clinical' (presence of genital lesions) or 'subclinical" (no genital lesions). The total shedding rate was defined for each participant as the percentage of all days (clinical and subclinical) on treatment during which shedding was detected by PCR. Genital/anal-rectal swabs was collected daily during each entire 60-day treatment period of each period and the washout period.
Time Frame: Up to Day 60 of each treatment period (up to 160 days)
Population: ITTC population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | VALTREX 1 g Once Daily | Placebo
Number analyzed (Participants) | 56 | 56
Percentage of days | 1.5 (5.2) | 5.5 (9.2)
Statistical Analysis 1: Comparison: VALTREX 1 g Once Daily vs Placebo; Test type: Superiority or Other; p < 0.001, Nonparametric tests-Wilcoxon Rank Sum

3. Secondary Outcome: Number of Participants With no Shedding
Description: The number of participants with no shedding was defined as the number of participants with no HSV-2 shedding detected by PCR divided by the total number of participants with PCR data. During each 60-day treatment period and during washout, swabs were collected daily from the genital/anal-rectal area for HSV-2 detection by PCR. During an outbreak, lesion swabs were also collected for HSV-2 detection by PCR. For each participant, each study day was classified by PCR as 'shedding' or 'no shedding'; additionally each day was classified as 'clinical' (presence of genital lesions) or 'subclinical" (no genital lesions).
Time Frame: Up to Day 60 of each treatment period (up to 160 days)
Population: ITTC population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | VALTREX 1 g Once Daily | Placebo
Number analyzed (Participants) | 56 | 56
Participants
  No Shedding | 47 | 30
  Shedding | 9 | 26
Statistical Analysis 1: Comparison: VALTREX 1 g Once Daily vs Placebo; Test type: Superiority or Other; p < 0.001, Prescott's method

4. Secondary Outcome: Mean Log HSV-2 DNA Copy Number Per Day on Days With Subclinical Shedding
Description: The subclinical shedding rate was defined for each participant as the total number of subclinical days on treatment during which shedding was detected by PCR. Average log HSV-2 DNA copy number per day on days with subclinical shedding was defined as the daily maximum HSV-2 DNA copy number was log transformed and averaged over all subclinical shedding days. During each 60-day treatment period and during washout, swabs were collected daily from the genital/anal-rectal area for HSV-2 detection by PCR. During an outbreak, lesion swabs were also collected for HSV-2 detection by PCR. For each participant, each study day was classified by PCR as 'shedding' or 'no shedding'; additionally each day was classified as 'clinical' (presence of genital lesions) or 'subclinical" (no genital lesions).
Time Frame: Up to Day 60 of each treatment period (up to 160 days)
Population: ITTC population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: DNA copies per day
Arm/Group | VALTREX 1 g Once Daily | Placebo
Number analyzed (Participants) | 5 | 5
DNA copies per day | 4.5 (0.9) | 4.6 (0.4)
Statistical Analysis 1: Comparison: VALTREX 1 g Once Daily vs Placebo; Test type: Superiority or Other; p = 0.800, Nonparametric tests-Wilcoxon Rank Sum

5. Secondary Outcome: Mean Log HSV-2 DNA Copy Number Per Day on Days With Total Shedding
Description: The total shedding rate was defined for each participant as the total number of all days (clinical and subclinical) on treatment during which shedding was detected by PCR. Average log HSV-2 DNA copy number per day on days with total shedding (clinical and subclinical) was defined as the daily maximum HSV-2 DNA copy number was log transformed and averaged over all shedding days. During each 60-day treatment period and during washout, swabs were collected daily from the genital/anal-rectal area for HSV-2 detection by PCR. During an outbreak, lesion swabs were also collected for HSV-2 detection by PCR. For each participant, each study day was classified by PCR as 'shedding' or 'no shedding'; additionally each day was classified as 'clinical' (presence of genital lesions) or 'subclinical" (no genital lesions).
Time Frame: Up to Day 60 of each treatment period (up to 160 days)
Population: ITTC population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: DNA copies per day
Arm/Group | VALTREX 1 g Once Daily | Placebo
Number analyzed (Participants) | 7 | 7
DNA copies per day | 4.5 (0.9) | 5.2 (1.2)
Statistical Analysis 1: Comparison: VALTREX 1 g Once Daily vs Placebo; Test type: Superiority or Other; p = 0.229, Nonparametric tests-Wilcoxon Rank Sum

6. Secondary Outcome: Percent Overall Study Population Who Have Recognized Clinical Signs/Symptoms of Genital Herpes Infection During the Study
Description: Participants who have recognized clinical signs/symptoms of genital herpes infection during the study. Participants were educated on recognizing signs and symptoms of genital herpes infection at the screening/randomization visit. Genital examinations was conducted at the randomization and genital herpes outbreak visits.
Time Frame: Up to Day 60 of each treatment period (up to 160 days)
Population: ITTC population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | VALTREX 1 g Once Daily | Placebo
Number analyzed (Participants) | 56 | 56
Percentage of participants
  No Signs/Symptoms | 88 | 77
  Signs/symptoms Present | 13 | 23
Statistical Analysis 1: Comparison: VALTREX 1 g Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0331, Prescott's method

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAE) were reported through out the study (up to 160 days)
Description: The ITTE population was used.
Arm/Group | Valtrex 1 g Once Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/65 | 1/63
Other Adverse Events (participants affected / at risk) | 29/65 | 42/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valtrex 1 g Once Daily (N=65) | Placebo (N=63)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valtrex 1 g Once Daily (N=65) | Placebo (N=63)
Upper respiratory tract infection (Infections and infestations) | 2 | 8
Nasopharyngitis (Infections and infestations) | 2 | 5
Vaginitis bacterial (Infections and infestations) | 1 | 3
Folliculitis (Infections and infestations) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 0 | 3
Stomach discomfort (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Oral soft tissue disorder (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 4
Dizziness (Nervous system disorders) | 4 | 1
Migraine (Nervous system disorders) | 2 | 1
Tension headache (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Failure of implant (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood urine present (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0
Metamyelocyte count increased (Investigations) | 1 | 0
Myelocyte count increased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.